CLINICAL TRIAL: NCT04833374
Title: Effect and Security of Steroids Therapy for Patients of IgA Nephropathy With Crescents : A Prospective, Randomized, Controlled, Multi-Center Clinical Trial.
Brief Title: Steroids Therapy in IgA Nephropathy With Crescents
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010PY (2020) -51
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; crescent; steroid; proteinuria; eGFR
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1-2-3 Group (Experimental): Patients in 1-2-3Group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-2nd-3rd month, then oral prednisone 0.5mg/kg/d on alternate days for 6 months.
  Interventions: Drug: Methylprednisolone
- 1-3-5 Group (Active Comparator): Patients in 1-3-5 Group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-3rd-5th month ,then oral prednisone 0.5mg/kg/d on alternate days for 6 months.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Patients will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-2nd-3rd or 1st-3rd-5th month, then oral prednisone 0.5mg/kg/d on alternate days for 6 months.
  Other Names: Prednisone

SUMMARY:
This prospective, randomized, controlled, multi-center clinical trial will evaluate the effect and security of steroids therapy for patients of IgA nephropathy with crescents.

DETAILED DESCRIPTION:
It has been reported that for urinary protein excretion that is persistently more than 1g/24h and eGFR>50ml/min/1.73m2 in IgA nephropathy(IgAN), the KDIGO guidelines suggest a 6-month course of glucocorticoids. The famous study by Pozzi C has proved that for patients of IgAN with proteinuria of 1.0-3.5g/24h and serum creatinine concentrations of 133 umol/L or less, a 6-month course of steroid treatment(1g/d methylprednisolone intravenously for 3 consecutive days, with the course repeated 2 months and 4 months later,then oral prednisone 0.5mg/kg/d on alternate days for 6 months) could significantly reduce proteinuria and protect against renal function deterioration in IgAN. However, according to Oxford classification, crescents in IgAN would effect the prognosis.This will be a prospective, randomized, controlled, multi-center study. Patients in treatment group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-2nd-3rd month ,then oral prednisone 0.5mg/kg/d on alternate days. Patients in control group will receive 0.5g/d methylprednisolone intravenously for 3 consecutive days in the 1st-3rd-5th month ,then oral prednisone 0.5mg/kg/d on alternate days. After followed-up for 6 months, the curative effect of steroid therapy on proteinuria and the progression of IgAN will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14~65 years, regardless of gender
2. Clinical evaluation and renal biopsy diagnostic for IgA nephropathy, presenting with crescents.
3. Average urinary protein excretion of 0.3~3.5g/24h on two successive examinations.
4. eGFR≥30 ml/min/1.73m2.
5. Willingness to sign an informed consent.

Exclusion Criteria:

1. Secondary IgAN such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B-associated nephritis, etc.
2. Rapidly progressive nephritic syndrome (crescent formation≥50%).
3. Acute renal failure, including rapidly progressive IgAN.
4. Current or recent (within 30 days) exposure to high-dose of steroids or immunosuppressive therapy (CTX、MMF、CsA、FK506).
5. Date of renal biopsy exceeds more than 30 days.
6. Cirrhosis, chronic active liver disease, and serious liver function damage.
7. History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease).
8. Any Active systemic infection or history of serious infection within one month.
9. Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure , chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases).
10. Active tuberculosis
11. Malignant hypertension that is difficult to be controlled by oral drugs.
12. Known allergy, contraindication or intolerance to the steroids.
13. Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception.
14. Malignant tumors.
15. Excessive drinking or drug abuse.
16. Mental aberrations.
17. Current or recent (within 30 days) exposure to any other investigational drugs.
18. Current use of RAS inhibitors needs to be eluted for at least 1 week before participating in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission of proteinuria | 6 months
  Proteinuria<0.3g/24h and stable renal function

SECONDARY OUTCOMES:
Partial remission of proteinuria | 6 months
  Proteinuria decline>50%, serum albumin>30g/L and stable renal function
Deterioration of renal function | 6 months
  The longitudinal decline of eGFR, serum creatinine arise>50%, or eGFR decline>25%, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pozzi C, Bolasco PG, Fogazzi GB, Andrulli S, Altieri P, Ponticelli C, Locatelli F. Corticosteroids in IgA nephropathy: a randomised controlled trial. Lancet. 1999 Mar 13;353(9156):883-7. doi: 10.1016/s0140-6736(98)03563-6. PMID 10093981
- [Result] Pozzi C, Andrulli S, Del Vecchio L, Melis P, Fogazzi GB, Altieri P, Ponticelli C, Locatelli F. Corticosteroid effectiveness in IgA nephropathy: long-term results of a randomized, controlled trial. J Am Soc Nephrol. 2004 Jan;15(1):157-63. doi: 10.1097/01.asn.0000103869.08096.4f. PMID 14694168
- [Result] Wyatt RJ, Julian BA. IgA nephropathy. N Engl J Med. 2013 Jun 20;368(25):2402-14. doi: 10.1056/NEJMra1206793. No abstract available. PMID 23782179
- [Result] Trimarchi H, Barratt J, Cattran DC, Cook HT, Coppo R, Haas M, Liu ZH, Roberts IS, Yuzawa Y, Zhang H, Feehally J; IgAN Classification Working Group of the International IgA Nephropathy Network and the Renal Pathology Society; Conference Participants. Oxford Classification of IgA nephropathy 2016: an update from the IgA Nephropathy Classification Working Group. Kidney Int. 2017 May;91(5):1014-1021. doi: 10.1016/j.kint.2017.02.003. Epub 2017 Mar 22. PMID 28341274
- [Result] Hotta O, Furuta T, Chiba S, Tomioka S, Taguma Y. Regression of IgA nephropathy: a repeat biopsy study. Am J Kidney Dis. 2002 Mar;39(3):493-502. doi: 10.1053/ajkd.2002.31399. PMID 11877568
- [Result] Shoji T, Nakanishi I, Suzuki A, Hayashi T, Togawa M, Okada N, Imai E, Hori M, Tsubakihara Y. Early treatment with corticosteroids ameliorates proteinuria, proliferative lesions, and mesangial phenotypic modulation in adult diffuse proliferative IgA nephropathy. Am J Kidney Dis. 2000 Feb;35(2):194-201. doi: 10.1016/s0272-6386(00)70326-x. PMID 10676716
- [Result] Rauen T, Eitner F, Fitzner C, Sommerer C, Zeier M, Otte B, Panzer U, Peters H, Benck U, Mertens PR, Kuhlmann U, Witzke O, Gross O, Vielhauer V, Mann JF, Hilgers RD, Floege J; STOP-IgAN Investigators. Intensive Supportive Care plus Immunosuppression in IgA Nephropathy. N Engl J Med. 2015 Dec 3;373(23):2225-36. doi: 10.1056/NEJMoa1415463. PMID 26630142
- [Result] Lv J, Zhang H, Wong MG, Jardine MJ, Hladunewich M, Jha V, Monaghan H, Zhao M, Barbour S, Reich H, Cattran D, Glassock R, Levin A, Wheeler D, Woodward M, Billot L, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Wang HY, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):432-442. doi: 10.1001/jama.2017.9362. PMID 28763548
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363